CLINICAL TRIAL: NCT06863831
Title: Yishen Qutong Granules vs. Simulant Combined With Neoadjuvant Chemoradiotherapy or Chemoimmunotherapy in the Treatment of Locally Advanced Esophageal Cancer: A Multicenter, Prospective, Double-Blind, Randomized Controlled Trial Protocol
Brief Title: A Multicenter Trial of YSQTG vs. Simulated Agents With Neoadjuvant Chemoradiotherapy or Chemoimmunotherapy for EC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: China-Japan Friendship Hospital (Other); Shanxi Provincial Cancer Hospital (Unknown); Changzhi People's Hospital (Other); Yuncheng Central Hospital (Other); Jilin Provincial Tumor Hospital (Other); Liaoning Cancer Hospital & Institute (Other); Shanghai Chest Hospital (Other); The Affiliated Hospital of Qingdao University (Other); Zhejiang Cancer Hospital (Other); Henan Cancer Hospital (Other Government); The First Affiliated Hospital of Zhengzhou University (Other); Wuhan No.1 Hospital (Other); Anyang Tumor Hospital (Other); Chongqing University Cancer Hospital (Other); Mianyang Central Hospital (Other); The Second Affiliated Hospital of Harbin Medical University (Other); The First Hospital of Jilin University (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NCC4369; 2023YFC3503200 (Other Grant/Funding Number: China National Center for Biotechnology Development)
Record Dates: First submitted 2025-02-17; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Esophageal Squamous Cell Carcinoma (ESCC)
Keywords: Traditional Chinese Medicine; Western Medicine
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Chemoradiotherapy TCM Treatment Group (Experimental): On the basis of neoadjuvant concurrent chemoradiotherapy (primarily based on a combination of Paclitaxel/Albumin-bound Paclitaxel, Cisplatin, and Radiotherapy), 10g/bag of Yishen Qutong Granules, 1 sachet per time, Tid, the administration cycle is the same as that of neoadjuvant concurrent chemoradiotherapy
  Interventions: Drug: Yishen Qutong Granules
- Chemoradiotherapy TCM Simulant Group (Placebo Comparator): On the basis of neoadjuvant concurrent chemoradiotherapy (primarily based on a combination of Paclitaxel/Albumin-bound Paclitaxel, Cisplatin, and Radiotherapy), 10g/bag of Yishen Qutong Granules (Yishen Qutong Simulant Granules, 1/10 Yishen Qutong Granules), 1 sachet per time, Tid, the administration cycle is the same as that of neoadjuvant concurrent chemoradiotherapy
  Interventions: Drug: Yishen Qutong Simulant Granules
- Chemoimmunotherapy TCM Treatment Group (Experimental): Neoadjuvant chemotherapy combined with immune drug therapy (primarily based on a combination of Karelizumab, a Platinum-based drug, and either Albumin-bound Paclitaxel or Paclitaxel) based on the use of Yishen Qutong Granules, 10g/dose, Tid treatment, synchronized with immunotherapy and chemotherapy
  Interventions: Drug: Yishen Qutong Granules
- Chemoimmunotherapy TCM Simulant Group (Placebo Comparator): Neoadjuvant chemotherapy combined with immune drug therapy (primarily based on a combination of Karelizumab, a Platinum-based drug, and either Albumin-bound Paclitaxel or Paclitaxel) based on the use of Yishen Qutong Simulant granules (1/10 Yishen Qutong Granules), 10g/dose, Tid treatment, used in tandem with immunotherapy, chemotherapy
  Interventions: Drug: Yishen Qutong Simulant Granules

INTERVENTIONS:
Drug: Yishen Qutong Granules — The patent prescription of Professor Feng Li, the head of the Department of Traditional Chinese Medicine at the Cancer Hospital of the Chinese Academy of Medical Sciences.
  Other Names: YSQTG
  Arms: Chemoimmunotherapy TCM Treatment Group; Chemoradiotherapy TCM Treatment Group
Drug: Yishen Qutong Simulant Granules — Yishen Qutong Simulant Granules is a preparation with one-tenth the dosage of Yishen Qutong Granules.
  Other Names: YSQTSG
  Arms: Chemoimmunotherapy TCM Simulant Group; Chemoradiotherapy TCM Simulant Group

SUMMARY:
Esophageal cancer is a high - incidence cancer type in China, characterized by high incidence, high mortality, and low survival rates. Over 90% of esophageal cancer cases in China are squamous cell carcinoma, while in Western countries, approximately 80% are adenocarcinomas. Current international guidelines, including those of the NCCN and CSCO, are not entirely suitable for the diagnosis and treatment of esophageal cancer in the Chinese context. In recent years, although the 5 - year survival rate for esophageal cancer has improved, significant challenges remain, such as severe side effects during chemoradiotherapy and targeted - immunotherapy, decreased patient tolerance and quality of life, and even interruption of treatment.

To leverage the synergistic role of traditional Chinese medicine (TCM) in the treatment of major diseases, this study, which builds on previous research, is founded on the theory of "reinforcing healthy qi to strengthen the body, removing toxins, and resolving stasis." It aims to conduct a multicenter, randomized, controlled clinical trial of the TCM formula Yishen Qutong Granules, designed to reinforce healthy qi to strengthen the body and remove toxins, in combination with neoadjuvant concurrent therapy for locally advanced esophageal squamous cell carcinoma. The study will enroll 268 patients (1:1 ratio) with locally advanced esophageal squamous cell carcinoma (cTNM stage III - IVa) who are expected to undergo neoadjuvant concurrent therapy and are potentially resectable. On the basis of conventional Western medical treatment, the treatment group will be administered the patented TCM formula Yishen Qutong Granules orally, while the control group will receive a Yishen Qutong Simulated Granules orally.

The primary outcome measure will be the clinical benefit rate (CBR, CBR = CR + PR + SD), with secondary outcomes including pathological response rate (mPR), R0 resection rate, and TCM syndrome symptom score. The study aims to establish an objective evaluation system for the efficacy and safety of combined treatment based on the integration of disease and syndrome differentiation. It will also elucidate the mechanisms underlying the therapeutic effects of Yishen Qutong Granules.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled clinical trial. The objective is to verify the efficacy and safety of Yishen Qutong Granules, a traditional Chinese medicine (TCM) for reinforcing healthy qi to strengthen the body and remove toxins, in combination with neoadjuvant concurrent chemoradiotherapy or neoadjuvant concurrent chemoimmunotherapy for locally advanced esophageal cancer that is expected to be resectable.

Patients will be recruited from the Cancer Hospital of the Chinese Academy of Medical Sciences and other collaborating clinical units involved in this project. The study will include two cohorts:

1. Patients undergoing neoadjuvant concurrent chemoradiotherapy:

1. A total of 268 patients with locally advanced esophageal cancer who are expected to undergo neoadjuvant concurrent chemoradiotherapy will be recruited. They will be randomly assigned in a 1:1 ratio to the treatment group and the control group, with 134 patients in each group.
2. The treatment group will receive neoadjuvant concurrent chemoradiotherapy (radiotherapy + albumin-bound paclitaxel + cisplatin) and will be administered Yishen Qutong Granules concurrently with the chemoradiotherapy, at a dose of 10g per dose, three times daily (Tid).
3. The control group will receive neoadjuvant concurrent chemoradiotherapy combined with a placebo (1/10 the dose of Yishen Qutong Granules), with the same timing, dosage, and duration of administration.
4. The primary efficacy endpoint is the clinical benefit rate (CBR = CR + PR + SD) after neoadjuvant treatment.
5. Secondary endpoints include the pathological response rate (mPR), R0 resection rate, incidence of radiation esophagitis, pain levels caused by radiation esophagitis, and TCM syndrome symptom scores.
6. Follow-up will be conducted every three months for a total of eight times (over two years), during which the progression-free survival (PFS) of patients will be recorded.

2. Patients undergoing neoadjuvant chemotherapy combined with immunotherapy:

1. A total of 268 patients with locally advanced esophageal squamous cell carcinoma who are expected to undergo neoadjuvant chemoimmunotherapy will be recruited. They will be randomly assigned in a 1:1 ratio to the treatment group and the control group, with 134 patients in each group.
2. The treatment group will receive neoadjuvant chemotherapy combined with immunotherapy (PD1 immunotherapy + albumin-bound paclitaxel + cisplatin) and will be administered Yishen Qutong Granules concurrently, at a dose of 10g per dose, three times daily (Tid).
3. The control group will receive neoadjuvant chemotherapy combined with immunotherapy and a placebo (1/10 the dose of Yishen Qutong Granules), with the same timing, dosage, and duration of administration.
4. The primary efficacy endpoints are the clinical benefit rate (CBR = CR + PR + SD) and symptom scores after neoadjuvant treatment.
5. Secondary endpoints include the pathological response rate (mPR), R0 resection rate, TCM syndrome scores, changes in tongue and pulse, and Numeric Rating Scale (NRS) scores.
6. Follow-up will be conducted every three months for a total of eight times (over two years), during which the progression-free survival (PFS) of patients will be recorded.

Yishen Qutong Granules have been approved as an in-house preparation by the Beijing Municipal Drug Administration (Beijing Drug Preparation No. Z20200072000). The formula consists of the following ingredients: Rehmannia glutinosa (20 g), Drynaria fortunei (10 g), Oldenlandia diffusa (10 g), Scutellaria barbata (10 g), Pheretima aspergillum (10 g), Dioscorea opposita (15 g), Cornus officinalis (15 g), Moutan cortex (10 g), Alisma plantago-aquatica (10 g), and Poria cocos (10 g). In this formula, Rehmannia glutinosa serves as the principal herb, nourishing yin and kidney essence, and enriching marrow. Cornus officinalis and Dioscorea opposita act as secondary herbs, with the former nourishing liver and kidney and the latter benefiting spleen yin. Oldenlandia diffusa and Scutellaria barbata detoxify, remove blood stasis, relieve pain, and inhibit cancer, while Pheretima aspergillum resolves blood stasis, unblocks meridians, and alleviates pain. Alisma plantago-aquatica drains dampness and purges turbidity, Moutan cortex clears fire and promotes blood circulation to remove blood stasis, and Poria cocos drains dampness from the spleen, all serving as adjuvant herbs. Drynaria fortunei, acting as a guiding herb, tonifies kidney, strengthens bones, and directs the other herbs to the affected area. Together, these herbs work synergistically to tonify the kidney, support healthy qi, resolve blood stasis, disperse nodules, detoxify, and relieve pain.

The Yishen Qutong Granules (Yishen Gu Kang Formula) were granted a patent prescription in 2017 (Patent No.: ZL201310582907.9). In 2020, the research team completed preclinical pharmaceutical studies and obtained approval for the in-house preparation (Beijing Drug Preparation No. Z20200072000). In September 2022, the technology was successfully transferred for a value of 20 million yuan, and the related achievements were awarded the Second Prize of the Beijing Science and Technology Progress Award in the same year. A total of 13 clinical and basic research projects have been conducted around the Yishen Gu Kang Formula, which has also been included in three guidelines, such as the "Guidelines for Integrated Traditional Chinese and Western Medicine Diagnosis and Treatment of Cancer Pain" by the China Association of Chinese Medicine. The preparation process and quality control standards of Yishen Qutong Granules were established by the Department of Pharmacy at the Cancer Hospital, Chinese Academy of Medical Sciences.

Sample Size Calculation

1. Chemoradiotherapy Group: The clinical benefit rate (CBR), defined as the proportion of patients achieving complete response (CR), partial response (PR), or stable disease (SD), was selected as the primary endpoint. Based on literature review and preliminary results of Yishen Qutong Granules, the estimated CBR for the treatment group was 0.88, while that for the neoadjuvant concurrent chemoradiotherapy group (paclitaxel + platinum-based chemotherapy with radiotherapy) was 0.73. With a two-sided α of 0.05 (one-sided α = 0.025) and a 1:1 allocation ratio between the treatment and control groups, the sample size was calculated using PASS software. The results indicated that 122 participants were required for each group. Accounting for a 10% dropout rate due to loss to follow-up or refusal, the final sample size was determined to be at least 134 participants per group, totaling 268 participants.
2. Chemoimmunotherapy Group: The primary efficacy endpoints included the clinical benefit rate (CBR) after neoadjuvant therapy and symptom improvement scores, with the latter used for sample size calculation. Based on literature review and preliminary data from Yishen Qutong Granules, the estimated symptom improvement rate was 0.799 for the treatment group and 0.6 for the control group. A non-inferiority margin of 0 (control group minus treatment group) was set, with a one-sided α of 0.025 and a β of 0.1. With a 1:1 allocation ratio, the calculated sample size was 107 participants per group, totaling 214 participants. Considering a 20% dropout rate, the final sample size was adjusted to 268 participants, with 134 participants in each group.

In this study, the following categorical variables were described using frequencies or percentages, and comparisons between groups were performed using the chi-square test or Fisher's exact test:

1. Clinical Benefit Rate (CBR): Defined as the percentage of evaluable cases achieving complete response (CR), partial response (PR), or stable disease (SD) after treatment.
2. Major Pathological Response (mPR): Defined as the proportion of patients with ≤10% viable tumor cells in the resected tissue specimens following neoadjuvant therapy.
3. R0 Resection Rate: Refers to the percentage of cases where the tumor was completely removed with no residual cancer cells detected at the surgical margins.
4. Incidence of Radiation Esophagitis: Defined as the proportion of enrolled patients diagnosed with radiation esophagitis, confirmed through medical history, symptoms, esophageal barium X-ray, and endoscopy.
5. Safety Indicators: Including routine blood, urine, and stool tests, liver and kidney function tests, and electrocardiogram results, analyzed statistically based on the presence or absence of abnormalities.

For continuous variables in this study, the Shapiro-Wilk test was used to assess normality. If the data followed a normal distribution, they were expressed as mean ± standard deviation, and comparisons between two groups were conducted using the independent samples t-test, while comparisons among multiple groups were performed using one-way ANOVA. If the data did not follow a normal distribution, they were expressed as median (interquartile range), and comparisons between two groups were conducted using the Mann-Whitney U test, while comparisons among multiple groups were performed using the Kruskal-Wallis rank-sum test. The continuous variables included:

1. Quality of Life (QLQ-C30) Score: Assessed using the EORTC Quality of Life Questionnaire Core 30 (QLQ-C30) to evaluate patients' quality of life.
2. Symptom Scores After Neoadjuvant Therapy: Comprising the sum of patient-reported symptom improvement scores and scores for tongue and pulse condition improvements.
3. Traditional Chinese Medicine (TCM) Syndrome Scores: Including the sum of scores for kidney deficiency syndrome and blood stasis-toxicity syndrome.
4. Progression-Free Survival (PFS): Defined as the time from randomization to tumor progression or death, with differences in PFS between groups compared using the Log-rank test.

All statistical analyses were performed using R software (version 4.0.3). Two-sided tests were applied, and a P-value <0.05 was considered statistically significant, with a significance level of α=0.05.

Quality Control and Assurance

1. The National Cancer Center/Cancer Hospital of the Chinese Academy of Medical Sciences serves as the leading and implementing institution, establishing a comprehensive organizational management system to ensure the successful completion of the project. The Quality Control Office is located within the Department of Cancer Prevention and Control at the National Cancer Center, overseen by Director Yawei Zhang, a project member and former tenured associate professor at the Yale School of Public Health, who was also selected under the Ministry of Science and Technology's "Thousand Talents Plan." Director Zhang is responsible for overall quality control and supervision. The project has designated one full-time project manager and one assistant to coordinate research activities and ensure the project's progress. They strictly adhere to the project requirements, comply with the management of the overarching project administration and the leading institution, submit regular progress reports, and promptly report any significant issues encountered during implementation.
2. A Project Management Office and an Advisory Committee composed of experts will be established. The Project Management Office, consisting of the principal investigator and full-time project managers, will handle daily operations, including monitoring and supervising the implementation of tasks across participating institutions. The Advisory Committee, organized by the principal investigator, will include technical, economic, and management experts in the field of esophageal cancer collaborative therapy. This committee will provide consultation on research protocols and technical issues, objectively evaluate the prospects of proposed research activities, offer recommendations, and ensure scientific rigor and feasibility through academic decision-making and quality oversight. Regular project coordination meetings will be held to determine the overall plan and technical strategies. In the event of major issues, the leading institution and the principal investigator will coordinate with the Advisory Committee to develop timely solutions and ensure corrective actions are implemented by relevant units, thereby guaranteeing the project's smooth progression.

Quality Assurance Plan: We will conduct regular data audits that encompass both automated data validation and manual review processes. The automated validation will utilize specialized software designed to assess data consistency and completeness, ensuring that all entered data adheres to predefined formats and ranges. Furthermore, annual on-site audits will be scheduled by an independent third-party entity to verify the compliance of data collection and processing procedures. Any discrepancies or errors identified will be documented, and corrective actions will be implemented promptly.

Data Checks: All data inputs will undergo a two-tier verification process. Initially, an automated system will perform a preliminary check based on predefined criteria such as data range, format, and logical relationships to identify potential errors or inconsistencies. Subsequently, research team members will conduct a manual review focusing on data flagged by the automated system and randomly selected additional data entries to ensure the accuracy and reliability of the data.

Source Data Verification: To ensure the accuracy of source data, we will implement a rigorous source data verification procedure. This involves comparing the data in the registry with the original data sources, such as medical records and laboratory reports. We will employ an electronic data capture system to minimize data entry errors and conduct regular checks for data consistency. Moreover, a 100% source data verification will be performed for key variables to guarantee the representativeness and accuracy of the data.

Data Dictionary: Patient ages will be extracted from electronic health records and encoded using WHO standards. All laboratory results will be retrieved from the central laboratory database and encoded according to MedDRA standards. The data dictionary will provide clear guidelines for each variable, ensuring data consistency and comparability.

Standard Operating Procedures (SOPs): We will establish Standard Operating Procedures (SOPs) for all critical operations within the study, including patient recruitment, data collection, data management, data analysis, and adverse event reporting. Each SOP will detail the steps to be taken, the responsible parties, and the timelines, ensuring consistency and reproducibility in all operations. For instance, the patient recruitment SOP will outline the recruitment process, screening criteria, and the informed consent procedure. The data collection SOP will specify the format and timing of data entry, as well as measures for data quality control.

ELIGIBILITY:
Inclusion Criteria:

1. Patients met the diagnostic criteria of expected resectable stage III-IVa esophageal cancer, and esophageal squamous cell carcinoma was confirmed by pathology. The diagnostic criteria refered to the guidelines for the diagnosis and treatment of esophageal cancer (2018 edition). Staging criteria: UICC/AJCC TNM staging system (8th edition, 2017) was used.
2. patients had not received previous treatment and planned to receive neoadjuvant simultaneous radiotherapy (radiotherapy + platinum in combination with albumin-paclitaxel), or proposed neoadjuvant chemotherapy in combination with immunopharmaceuticals (Immunotherapy reference 2024 CSCO Esophageal Cancer Diagnosis and Treatment Guidelines + platinum in combination with albumin-paclitaxel)
3. In accordance with the syndrome type of positive deficiency and toxin stasis (kidney deficiency and deficiency syndrome + blood stasis and toxin stagnation syndrome), that is, at least one main symptom + two secondary symptoms in each syndrome scale;
4. Karnofsky Performance Scale (KPS) ≥70; (5)18 ≤ age ≤ 80 ;

(6) Patients who agreeed to participate in this study and sign the informed consent form.

Exclusion Criteria:

1. ①Yishen Qutong Granules Comparison Simulator Cooperative Neoadjuvant Synchronized Radiotherapy Group: those who have contraindications to radiotherapy such as esophageal fistula or those who are allergic to chemotherapeutic drugs; ②Yishen Qutong Granules Comparison Simulator Cooperative Neoadjuvant Chemotherapy Combined with Immunotherapy Drugs Group: those who have contraindications to chemotherapy and immunotherapy or those who are allergic to the drugs;
2. patients with a history of other tumors, cardiovascular and cerebrovascular diseases, liver and kidney function damage, hematopoietic system diseases, and other serious diseases;
3. patients with mental disorders;
4. patients during pregnancy and lactation;
5. patients allergic to traditional Chinese medicine used in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 536 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
clinical benefit rate (CBR) | Assessed after completion of neoadjuvant therapy (2-4 cycles) and post-surgery, typically within 2-5 months after enrollment.
  clinical benefit rate, CBR=(CR+PR+SD)
Symptom Score | Assessed at the end of each treatment cycle (each cycle is 28 days), up to 5 cycles.
  Assess the symptom scores of esophageal squamous cell carcinoma using a questionnaire.
  Esophageal Cancer Obstruction and Dysphagia Symptom Score:
  0: No obstruction, does not affect eating at all
  1. Very mild sensation of obstruction, does not affect eating
  2. Mild obstruction, does not affect eating
  3. Mild obstruction but occasionally increased sensation of obstruction, very mildly affects eating, does not affect intake of liquids
  4. Mild obstruction, mildly affects eating
  5. Mild obstruction but occasionally increased sensation of obstruction, affects eating, including liquids
  6. Moderate obstruction, affects eating, including liquids
  7. Moderate obstruction and occasionally increased sensation of obstruction, can only swallow liquids
  8. Severe obstruction, can only consume very thin liquids
  9. Severe obstruction, can only drink water
  10. Complete obstruction

SECONDARY OUTCOMES:
mPR resection rate | At the end of the surgery
  The mPR resection rate is evaluated through postoperative pathology.
R0 resection rate | At the end of the surgery
  R0 resection rate is evaluated through postoperative pathology.
QLQ-C30 scale point | Assessed at the end of each treatment cycle (each cycle is 28 days), up to 5 cycles.
  Outcome Measure: Quality of Life assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30).
  Description: The EORTC QLQ-C30 is a 30-item questionnaire evaluating cancer patients' quality of life across multiple dimensions, including physical, emotional, cognitive, and social functioning, as well as symptom burden (e.g., fatigue, pain, nausea). Scores range from 0 to 100, with higher scores in functional scales and global health status indicating better quality of life, and higher scores in symptom scales indicating worse symptoms.
  Time Frame: Assessed at baseline, after each treatment cycle (each cycle is 28 days), and at the end of treatment.
The NRS degree of pain caused by radiation esophagitis | Assessed at the end of each treatment cycle (each cycle is 28 days), up to 5 cycles.
  The Numeric Rating Scale (NRS) for pain is a simple and straightforward tool for assessing pain levels. It consists of 11 numbers ranging from 0 to 10, allowing patients to select the number that best represents the intensity of their pain, with 0 indicating no pain and 10 indicating the most severe pain. Pain often comes with an impact on sleep quality. On this NRS scale, 0-3 represents no effect on sleep, 4-6 indicates a mild effect on sleep, and 7-10 signifies an inability to sleep or being awakened by pain. Patients choose a number between 0 and 10 to represent their level of pain intensity. The higher the number, the more severe the pain.
Evaluation of Syndrome and Symptom Points of Traditional Chinese Medicine | Assessed at the end of each treatment cycle (each cycle is 28 days), up to 5 cycles.
  Outcome Measure: Traditional Chinese Medicine (TCM) Syndrome Score. Description: The TCM Syndrome Score evaluates the severity of symptoms related to nodule accumulation, localized pain, tongue appearance, lumbar debility, and fatigue. Each symptom is scored from 0 to 6, with higher scores indicating more severe symptoms. The total score is the sum of individual symptom scores, reflecting the overall severity of TCM syndromes.
  Time Frame: Assessed at baseline, after each treatment cycle (each cycle is 28 days), and at the end of treatment.
Progression free survival (PFS) | After the completion of neoadjuvant concurrent therapy, patients will be followed up every 3 months for a total of 8 times (over 2 years), and their progression-free survival (PFS) will be recorded.
  Progression-Free Survival (PFS) is a commonly used endpoint in oncology clinical research, used to assess the time from the start of treatment to disease progression or death.
pathological complete response rate (pCR) | Assessed by surgical pathology within 10 days after surgery.
  Pathological complete response (pCR) refers to the absence of viable tumor cells in the resected tumor tissue and regional lymph nodes.
KPS score | Assessed at the end of each treatment cycle (each cycle is 28 days), up to 5 cycles.
  The Karnofsky Performance Status (KPS) score is a tool used to assess a patient's functional status and quality of life, and it is widely applied in the fields of oncology and palliative care.
  100: Fully active, able to carry on all pre-disease activities without restriction.
  90: Capable of normal activity with minor signs or symptoms of disease. 80: Normal activity with effort; some signs or symptoms of disease. 70: Cares for self but unable to carry on normal activity or active work. 60: Requires occasional assistance but is able to care for most of their personal needs.
  50: Requires considerable assistance and frequent medical care. 40: Disabled; requires special care and assistance. 30: Severely disabled; hospitalization is indicated although death not imminent.
  20: Very sick; hospitalization necessary; active treatment may be indicated. 10: Moribund; fatal processes progressing rapidly. 0: Dead.
Changes of the tongue | Assessed at the end of each treatment cycle (each cycle is 28 days), up to 5 cycles.
  Detect changes in the patient's tongue using a tongue detector.
Changes of the pulse | Assessed at the end of each treatment cycle (each cycle is 28 days), up to 5 cycles.
  Detect changes in the patient's pulse using a pulse detector.

CONTACTS AND LOCATIONS:
Overall Officials: Li Feng, Ph.D., Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences/Peking Union Medical College, Beijing, Chaoyang, China

IPD SHARING:
Plan to Share IPD: No
The project involves some patents that will not be disclosed at this time.

REFERENCES:
- [Background] Deboever N, Jones CM, Yamashita K, Ajani JA, Hofstetter WL. Advances in diagnosis and management of cancer of the esophagus. BMJ. 2024 Jun 3;385:e074962. doi: 10.1136/bmj-2023-074962. PMID 38830686
- [Background] DaSilva LL, Aguiar PN Jr, de Lima Lopes G. Immunotherapy for Advanced Esophageal Squamous Cell Carcinoma-Renewed Enthusiasm and a Lingering Challenge. JAMA Oncol. 2021 Nov 1;7(11):1613-1614. doi: 10.1001/jamaoncol.2021.4410. No abstract available. PMID 34519775
- [Background] Ying J, Zhang M, Qiu X, Lu Y. The potential of herb medicines in the treatment of esophageal cancer. Biomed Pharmacother. 2018 Jul;103:381-390. doi: 10.1016/j.biopha.2018.04.088. Epub 2018 Apr 24. PMID 29674273
- [Background] Zhang YS, Shen Q, Li J. Traditional Chinese medicine targeting apoptotic mechanisms for esophageal cancer therapy. Acta Pharmacol Sin. 2016 Mar;37(3):295-302. doi: 10.1038/aps.2015.116. Epub 2015 Dec 28. PMID 26707140
- [Background] The Lancet. GLOBOCAN 2018: counting the toll of cancer. Lancet. 2018 Sep 22;392(10152):985. doi: 10.1016/S0140-6736(18)32252-9. Epub 2018 Sep 20. No abstract available. PMID 30264708
- [Background] Conway E, Wu H, Tian L. Overview of Risk Factors for Esophageal Squamous Cell Carcinoma in China. Cancers (Basel). 2023 Nov 27;15(23):5604. doi: 10.3390/cancers15235604. PMID 38067307
- [Background] Morgan E, Soerjomataram I, Rumgay H, Coleman HG, Thrift AP, Vignat J, Laversanne M, Ferlay J, Arnold M. The Global Landscape of Esophageal Squamous Cell Carcinoma and Esophageal Adenocarcinoma Incidence and Mortality in 2020 and Projections to 2040: New Estimates From GLOBOCAN 2020. Gastroenterology. 2022 Sep;163(3):649-658.e2. doi: 10.1053/j.gastro.2022.05.054. Epub 2022 Jun 4. PMID 35671803
- [Background] Liu J, Yang Y, Liu Z, Fu X, Cai X, Li H, Zhu L, Shen Y, Zhang H, Sun Y, Chen H, Yu B, Zhang R, Shao J, Zhang M, Li Z. Multicenter, single-arm, phase II trial of camrelizumab and chemotherapy as neoadjuvant treatment for locally advanced esophageal squamous cell carcinoma. J Immunother Cancer. 2022 Mar;10(3):e004291. doi: 10.1136/jitc-2021-004291. PMID 35338088
- [Background] Lu Z, Wang J, Shu Y, Liu L, Kong L, Yang L, Wang B, Sun G, Ji Y, Cao G, Liu H, Cui T, Li N, Qiu W, Li G, Hou X, Luo H, Xue L, Zhang Y, Yue W, Liu Z, Wang X, Gao S, Pan Y, Galais MP, Zaanan A, Ma Z, Li H, Wang Y, Shen L; ORIENT-15 study group. Sintilimab versus placebo in combination with chemotherapy as first line treatment for locally advanced or metastatic oesophageal squamous cell carcinoma (ORIENT-15): multicentre, randomised, double blind, phase 3 trial. BMJ. 2022 Apr 19;377:e068714. doi: 10.1136/bmj-2021-068714. PMID 35440464
- [Background] Luo H, Lu J, Bai Y, Mao T, Wang J, Fan Q, Zhang Y, Zhao K, Chen Z, Gao S, Li J, Fu Z, Gu K, Liu Z, Wu L, Zhang X, Feng J, Niu Z, Ba Y, Zhang H, Liu Y, Zhang L, Min X, Huang J, Cheng Y, Wang D, Shen Y, Yang Q, Zou J, Xu RH; ESCORT-1st Investigators. Effect of Camrelizumab vs Placebo Added to Chemotherapy on Survival and Progression-Free Survival in Patients With Advanced or Metastatic Esophageal Squamous Cell Carcinoma: The ESCORT-1st Randomized Clinical Trial. JAMA. 2021 Sep 14;326(10):916-925. doi: 10.1001/jama.2021.12836. PMID 34519801
- [Background] Yang H, Liu H, Chen Y, Zhu C, Fang W, Yu Z, Mao W, Xiang J, Han Y, Chen Z, Yang H, Wang J, Pang Q, Zheng X, Yang H, Li T, Zhang X, Li Q, Wang G, Chen B, Mao T, Kong M, Guo X, Lin T, Liu M, Fu J. Long-term Efficacy of Neoadjuvant Chemoradiotherapy Plus Surgery for the Treatment of Locally Advanced Esophageal Squamous Cell Carcinoma: The NEOCRTEC5010 Randomized Clinical Trial. JAMA Surg. 2021 Aug 1;156(8):721-729. doi: 10.1001/jamasurg.2021.2373. PMID 34160577
- [Background] Wang ZX, Cui C, Yao J, Zhang Y, Li M, Feng J, Yang S, Fan Y, Shi J, Zhang X, Shen L, Shu Y, Wang C, Dai T, Mao T, Chen L, Guo Z, Liu B, Pan H, Cang S, Jiang Y, Wang J, Ye M, Chen Z, Jiang D, Lin Q, Ren W, Wang J, Wu L, Xu Y, Miao Z, Sun M, Xie C, Liu Y, Wang Q, Zhao L, Li Q, Huang C, Jiang K, Yang K, Li D, Liu Y, Zhu Z, Chen R, Jia L, Li W, Liao W, Liu HX, Ma D, Ma J, Qin Y, Shi Z, Wei Q, Xiao K, Zhang Y, Zhang Y, Chen X, Dai G, He J, Li J, Li G, Liu Y, Liu Z, Yuan X, Zhang J, Fu Z, He Y, Ju F, Liu Z, Tang P, Wang T, Wang W, Zhang J, Luo X, Tang X, May R, Feng H, Yao S, Keegan P, Xu RH, Wang F. Toripalimab plus chemotherapy in treatment-naive, advanced esophageal squamous cell carcinoma (JUPITER-06): A multi-center phase 3 trial. Cancer Cell. 2022 Mar 14;40(3):277-288.e3. doi: 10.1016/j.ccell.2022.02.007. Epub 2022 Mar 3. PMID 35245446
- [Background] Obermannova R, Alsina M, Cervantes A, Leong T, Lordick F, Nilsson M, van Grieken NCT, Vogel A, Smyth EC; ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org. Oesophageal cancer: ESMO Clinical Practice Guideline for diagnosis, treatment and follow-up. Ann Oncol. 2022 Oct;33(10):992-1004. doi: 10.1016/j.annonc.2022.07.003. Epub 2022 Jul 29. No abstract available. PMID 35914638
- [Background] Ajani JA, D'Amico TA, Bentrem DJ, Cooke D, Corvera C, Das P, Enzinger PC, Enzler T, Farjah F, Gerdes H, Gibson M, Grierson P, Hofstetter WL, Ilson DH, Jalal S, Keswani RN, Kim S, Kleinberg LR, Klempner S, Lacy J, Licciardi F, Ly QP, Matkowskyj KA, McNamara M, Miller A, Mukherjee S, Mulcahy MF, Outlaw D, Perry KA, Pimiento J, Poultsides GA, Reznik S, Roses RE, Strong VE, Su S, Wang HL, Wiesner G, Willett CG, Yakoub D, Yoon H, McMillian NR, Pluchino LA. Esophageal and Esophagogastric Junction Cancers, Version 2.2023, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2023 Apr;21(4):393-422. doi: 10.6004/jnccn.2023.0019. PMID 37015332
- [Background] Yang H, Wang F, Hallemeier CL, Lerut T, Fu J. Oesophageal cancer. Lancet. 2024 Nov 16;404(10466):1991-2005. doi: 10.1016/S0140-6736(24)02226-8. PMID 39550174
- [Background] Qi L, Wang J, Hou S, Liu S, Zhang Q, Zhu S, Liu S, Zhang S. Unraveling the tumor microenvironment of esophageal squamous cell carcinoma through single-cell sequencing: A comprehensive review. Biochim Biophys Acta Rev Cancer. 2025 Feb;1880(1):189264. doi: 10.1016/j.bbcan.2025.189264. Epub 2025 Jan 11. PMID 39805342